CLINICAL TRIAL: NCT00621517
Title: Bupropion and Restless Legs Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: East Tennessee State University (Other)
Responsible Party: Principal Investigator, Max Bayard, Associate Professor of Family Medicine, East Tennessee State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ETSU-07-061f
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Results first posted 2012-04-05 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-02

CONDITIONS: Restless Legs Syndrome
Keywords: Restless Legs Syndrome; Bupropion
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will receive 150MG Bupropion nightly.
  Interventions: Drug: Bupropion
- 2 (Placebo Comparator): Participants will receive matching placebo capsule nightly.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bupropion — Partipants will receive 150 mg bupropion per night
  Other Names: Wellbutrin
  Arms: 1
Drug: Placebo — 1 capsule nightly for six weeks
  Arms: 2

SUMMARY:
The purpose of this study is to determine if bupropion will improve the symptoms of restless legs syndrome (RLS).

DETAILED DESCRIPTION:
Adult patients with moderate to severe RLS will be recruited for the study. Those on medications which treat RLS will be asked to discontinue the medications for two weeks prior to beginning the study. All participants will be screened with Beck Depression Inventory, International Restless Legs Syndrome Study Group (IRLSSG) severity scale, and Clinical Global Impression of Improvement (CGI-I) scale. An ordinal scale (i.e. rate symptoms from 1-8) will also be obtained. Participants will be randomized to a placebo or medication group. Those in the medication group will be given 150 mg of bupropion at night for six weeks. Others will receive similar-appearing placebo. Participants will be called at the end of weeks one, two, four and five to assess symptom severity based on IRLSSG scale, and to determine if they are experiencing any adverse effects. At three weeks and six weeks, participants will return to the clinic to complete all four of the initial forms, the Beck Depression Inventory, IRLSSG severity scale, ordinal scale, and CGI-I.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Restless Legs Syndrome
* Severity Scale score 15 or higher

Exclusion Criteria:

* History of seizures
* History of alcohol use greater than 2 drinks per day or occasional binges of 5 or more drinks per day
* Suicidal thoughts/ideations
* Inability to return for follow up appointments at 3 and 6 weeks
* Lack of access to telephone
* Eating disorder
* Age less than 18
* Pregnancy
* Unwillingness or inability to discontinue any RLS medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- East Tennessee State University, Johnson City, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupropion: Participants will receive 150MG Bupropion nightly.
- Placebo: Participants will receive matching placebo capsule nightly.
Period: Overall Study
Arm/Group | Bupropion | Placebo
Started | 29 | 31
Completed | 22 | 24
Not Completed | 7 | 7
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupropion | Placebo | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 25 | 52
  >=65 years | 2 | 6 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (12.9) | 50.5 (14.1) | 49.3 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 46
  Male | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 29 | 31 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change in International Restless Legs Syndrome Study Group (IRLSSG) Severity Scale.
Description: Scale ranges from 0 to 40 points with higher scores being associated with more severe symptoms of restless legs syndrome. There are 10 questions, with points of 0 to 4 per question. The change in IRLSSG score from baseline is recorded at three and six weeks.
Time Frame: Baseline, three weeks, and six weeks
Population: Intention to Treat
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Bupropion | Placebo
Number analyzed (Participants) | 29 | 31
points on a scale
  Change in IRLSSG score from baseline to 6 weeks | -10.4 (10.1) | -7.6 (7.1)
  Change in IRLSSG score from baseline to 3 weeks | -10.8 (10.0) | -6.0 (6.6)

2. Primary Outcome: Clinical Global Impression - Improvement Scale
Time Frame: three weeks and six weeks
Population: Once we started recruiting patients, we had decided not to do this outcome so this data was not obtained.
Arm/Group | Bupropion | Placebo
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Ordinal Scale (i.e., 1-8) of Symptom Severity
Time Frame: three weeks and six weeks
Population: Once we started recruiting patients, we had decided not to do this outcome so this data was not obtained.
Arm/Group | Bupropion | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Bupropion | Placebo
Serious Adverse Events (participants affected / at risk) | 1/29 | 0/31
Other Adverse Events (participants affected / at risk) | 1/29 | 2/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Bupropion (N=29) | Placebo (N=31)
miscarriage (Pregnancy, puerperium and perinatal conditions) | 1/22 | 0/24 — Pregnancy was an exclusion criterion; participant denied pregnancy initially. Following this event, criteria to avoid possibility of similar event were added.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupropion (N=29) | Placebo (N=31)
nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
Possible Type II error as we were unable to recruit our target of 100 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No